CLINICAL TRIAL: NCT07027670
Title: Pre-operative 5-Aminolevulinic Acid to Activate Haem Oxygenase to Improve Outcomes in Cardiac Surgery: A Dose Finding Study
Brief Title: Treatment With 5-AminoLEvuliNic Acid Before Cardiac Surgery
Acronym: TALEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: SBI Pharmaceuticals Co, Ltd. (Industry); Emerald Clinical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 280513
Record Dates: First submitted 2022-05-03; First posted 2025-06-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Surgical Procedures; Coronary Artery Bypass; Aortic Valve Disease; Mitral Valve Disease
Keywords: heme oxygenase; cardiopulmonary bypass; HO-1; aortic valve replacement; mitral valve surgery; 5-aminolevulinic acid; delta aminolevulinic acid; sodium ferrous citrate
MeSH Terms: conditions — Aortic Valve Disease | interventions — Aminolevulinic Acid; ferrous citrate

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation cohorts of 10 evaluable patients each (8 on active:2 on placebo) dosed twice daily (bd) with 5-ALA-SFC or placebo for three pre-operative days and once on the day of cardiac surgery. Up to 4 discrete dose levels are anticipated.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation will follow a sequential randomisation list prepared by the blinded trial statistician. As participants are randomised, they will be manually allocated the next available treatment kit (active or placebo) number from this list which will correspond to the randomisation number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 75 mg 5-ALA with 118 mg SFC bd (lowest/starting dose) for three days before surgery (n=8 patients)
  Interventions: Drug: 5-Aminolevulinic Acid hydrochloride (5-ALA); Drug: Sodium ferrous citrate (SFC)
- Cohort 2 (Experimental): 150 mg 5-ALA with 236 mg SFC or bd for three days before surgery (n=8 patients)
  Interventions: Drug: 5-Aminolevulinic Acid hydrochloride (5-ALA); Drug: Sodium ferrous citrate (SFC)
- Cohort 3 (Experimental): 225 mg 5-ALA with 354 mg SFC bd for three days before surgery (n=8 patients)
  Interventions: Drug: 5-Aminolevulinic Acid hydrochloride (5-ALA); Drug: Sodium ferrous citrate (SFC)
- Cohort 4 (Experimental): 300 mg 5-ALA with 472 mg SFC bd (maximum dose) for three days before surgery (n=8 patients)
  Interventions: Drug: 5-Aminolevulinic Acid hydrochloride (5-ALA); Drug: Sodium ferrous citrate (SFC)
- Placebo (Placebo Comparator): 2 patients in each cohort above will be allocated to placebo (n=8 patients in total across the study)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 5-Aminolevulinic Acid hydrochloride (5-ALA) — 5-ALA: supplied for oral administration as a dark green, opaque, size 0, hypromellose (HPMC) capsule containing drug alone at a dosage strength of 75mg (58.7mg as 5-ALA). There are no excipients.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Other: Placebo — Supplied for oral administration as a dark green, opaque, size 0, HPMC capsule containing 125mg lactose. The capsule shells are of non-animal origin, and are comprised of HPMC, titanium dioxide, and a copper complex of chlorophyllins.
  Arms: Placebo
Drug: Sodium ferrous citrate (SFC) — SFC: supplied for oral administration as a dark green, opaque, size 0, HPMC capsule containing drug alone at a dosage strength 118mg (12.5mg as Fe). There are no excipients.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4

SUMMARY:
TALEN is a prospective randomised double-blind placebo-controlled phase 2 study of 5-Aminolevulinic Acid with Sodium Ferrous Citrate (5-ALA-SFC) in adult patients undergoing cardiac surgery on cardiopulmonary bypass (CPB). TALEN aims to identify the optimal biological dose (OBD) of 5-ALA-SFC.

DETAILED DESCRIPTION:
TALEN is a prospective, randomised, double blind, placebo-controlled phase 2 study of 5-ALA-SFC administration in adults undergoing non-emergent cardiac surgery on CPB examining the potential of 5-ALA-SFC to induce haem oxygenase-1 (HO-1) as a novel cardio- and cyto-protective strategy for clinical benefit. 5-ALA is an amino acid found in several foods and a natural endogenous precursor in the synthesis of haem. Oral administration of 5-ALA-SFC has been shown to be safe and to induce a pharmacodynamic effect on the key effector, HO-1. TALEN is designed as a dose-finding trial with sequential dose cohorts, evaluating the safety, tolerability and PD response to 5-ALA-SFC to determine the optimum biological dose for further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for non-emergent cardiac surgery under CPB (including coronary artery bypass grafting, valve replacement, valve repair or a combination thereof)
* Signed informed consent
* Age ≥18 years
* Able and willing to comply with all study requirements

Exclusion Criteria:

* Female participants who are of childbearing potential who are either unable or unwilling to use highly effective contraception, or who are pregnant or breast feeding
* History of hypersensitivity to 5-ALA, SFC and/or porphyrins
* Acute or chronic types of porphyria
* Known genetic haemochromatosis or clinically significant iron overload
* History of clinically significant photosensitization
* Current long-term (> 3 months) use of amiodarone
* Concomitant use of hypericin extract (including St John's Wort) or concomitant therapeutic dose oral iron replacement
* Use of other investigational medical product(s) < 28 days prior to study or 5 half-lives, whichever is longer
* Cardiogenic shock/Low cardiac output syndrome requiring catecholamine infusion and/or mechanical circulatory support prior to induction of anaesthesia for cardiac surgery
* Recent acute myocardial infarction
* Cardiac surgery without cardiopulmonary bypass or induced fibrillating heart surgery
* Inadequate renal or liver function
* Any other condition which, in the opinion of the Investigator, makes the patient unsuitable for or may compromise their participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline HO-1 expression to time of cardiac surgery | Baseline at screening compared to post dose (measured within 12 hours of final dose, before cardiac surgery)
  Normalised HO-1 expression in peripheral blood
  •Safety: Occurrence of adverse events / laboratory safety events defined as dose-limiting toxicity (DLTs)
Number of Participants With Dose Limiting Toxicity | Up to 72 hours post-surgery

SECONDARY OUTCOMES:
Incidence of treatment related emergent AEs [safety and tolerability] | From time of administration of placebo or investigational medicinal product (IMP) (i.e. treatment-emergent AEs, TEAEs) to 72 hours post-operatively
  Treatment-related AEs assessed using CTCAE v5.0
Change from baseline HO activity to time of cardiac surgery | Baseline at screening compared to post dose (measured within 12 hours of final dose, before cardiac surgery)
  HO enzyme activity
Preliminary evaluation of the kinetics of peri-operative myocardial injury | Serial measurements until 72 hours after release of aortic cross clamping
  Cardiac troponin area under the curve for 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Arash Yavari, DPhil MRCP, Principal Investigator — University of Oxford
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No